CLINICAL TRIAL: NCT06995352
Title: Liposomal Bupivacaine Versus Continuous Peripheral Nerve Blocks for Analgesia Following Ankle Surgery: A Randomized, Observer and Participant Masked, Active Control, Non-Inferiority Study
Brief Title: Liposomal Bupivacaine Versus Continuous Peripheral Nerve Blocks for Analgesia Following Ankle Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Pacira Biosciences (Unknown)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LipoBupiv vs cPNB (Ankle)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Moderate-to-severely Painful Ankle Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, participant- and observer-masked, active-control study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All individuals will be masked to treatment group assignment with the exception of the investigational pharmacists who prepare the study medication and the investigators who are administering the single-injection peripheral nerve blocks and inserting the perineurial catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine (Experimental) (Experimental): Popliteal-sciatic nerve block: 10 mL of unencapsulated bupivacaine 0.375% and 10 mL of liposomal bupivacaine 1.33% (Exparel, Pacira BioSciences, Tampa, Florida) admixed within a 20 mL syringe.
  Adductor canal (saphenous) nerve block: 10 mL of unencapsulated bupivacaine 0.375% and 10 mL of liposomal bupivacaine 1.33% (Exparel, Pacira BioSciences, Tampa, Florida) admixed within a 20 mL syringe.
  Postoperative perineural infusion: Basal rate 5 mL/h; patient-controlled bolus of 4 mL; 30 minute lockout; and reservoir with normal saline (500 mL).
  Interventions: Drug: Popliteal nerve block including liposomal bupivacaine; Drug: Adductor canal nerve block including liposomal bupivacaine; Drug: Continuous popliteal nerve block with normal saline
- Unencapsulated Bupivacaine (Control) (Active Comparator): Popliteal-sciatic nerve block: 20 mL of unencapsulated bupivacaine 0.375% with epinephrine (1:400,000) within a 20 mL syringe.
  Adductor canal (saphenous) nerve block: Standard-of-Care Group: 20 mL of unencapsulated bupivacaine 0.375% with epinephrine (1:400,000) within a 20 mL syringe.
  Postoperative perineural infusion: Basal rate 5 mL/h; patient-controlled bolus of 4 mL; 30 minute lockout; and reservoir of unencapsulated bupivacaine 0.125% (500 mL).
  Interventions: Drug: Popliteal nerve block with exclusively unencapsulated bupivacaine; Drug: Adductor canal nerve block with exclusively unencapsulated bupivacaine; Drug: Continuous popliteal nerve block with unencapsulated bupivacaine

INTERVENTIONS:
Drug: Popliteal nerve block including liposomal bupivacaine — 10 mL of unencapsulated bupivacaine 0.375% and 10 mL of liposomal bupivacaine 1.33% (Exparel, Pacira BioSciences, Tampa, Florida) admixed within a 20 mL syringe.
  Arms: Liposomal Bupivacaine (Experimental)
Drug: Adductor canal nerve block including liposomal bupivacaine — 10 mL of unencapsulated bupivacaine 0.375% and 10 mL of liposomal bupivacaine 1.33% (Exparel, Pacira BioSciences, Tampa, Florida) admixed within a 20 mL syringe.
  Arms: Liposomal Bupivacaine (Experimental)
Drug: Continuous popliteal nerve block with normal saline — A perineurial infusion of normal saline (basal rate 5 mL/h; patient-controlled bolus of 4 mL; 30 minute lockout) with the reservoir (500 mL) and pump provided by the Investigational Drug Service and continued until postoperative day 3 or until the reservoir is exhausted.
  Arms: Liposomal Bupivacaine (Experimental)
Drug: Popliteal nerve block with exclusively unencapsulated bupivacaine — 20 mL of unencapsulated bupivacaine 0.375% with epinephrine (1:400,000) within a 20 mL syringe.
  Arms: Unencapsulated Bupivacaine (Control)
Drug: Adductor canal nerve block with exclusively unencapsulated bupivacaine — 20 mL of unencapsulated bupivacaine 0.375% with epinephrine (1:400,000) within a 20 mL syringe.
  Arms: Unencapsulated Bupivacaine (Control)
Drug: Continuous popliteal nerve block with unencapsulated bupivacaine — A perineurial infusion of unencapsulated bupivacaine 0.125% (basal rate 5 mL/h; patient-controlled bolus of 4 mL; 30 minute lockout) with the reservoir (500 mL) and pump provided by the Investigational Drug Service and continued until postoperative day 3 or until the reservoir is exhausted.
  Arms: Unencapsulated Bupivacaine (Control)

SUMMARY:
Postoperative pain remains undertreated. Opioids have well-known limitations for both individuals and society, and while single-injection peripheral nerve blocks with unencapsulated local anesthetic provide potent analgesia, their duration is measured in hours while post-surgical pain usually outlasts this duration. Continuous peripheral nerve blocks prolong analgesia but may possibly be replaced with liposomal bupivacaine with a reported duration of up to 72-96 hours (Schwartz. J Clin Anesth 2024). In comparison to continuous peripheral nerve blocks, liposomal bupivacaine eliminates a time-consuming catheter insertion as well as the risks of catheter dislodgement, localized infection, local anesthetic leakage, and infusion pump malfunction. Furthermore, liposomal bupivacaine significantly reduces the burden on both patients and healthcare providers as it does not require the use of a portable infusion pump, local anesthetic reservoir, or perineural catheter to be carried, managed, or eventually removed. Notably, the potential for local anesthetic-induced myotoxicity, and cardiac/neurologic toxicity is reduced or negated altogether. And the cost of liposome bupivacaine is less than the combined cost of a catheter set, insertion equipment, portable infusion pump, large reservoir of local anesthetic, and healthcare provider oversight.

Therefore, should a single injection of liposomal bupivacaine be demonstrated to provide at least non-inferior analgesia and opioid sparing as a continuous peripheral nerve block, it would be a far superior analgesic benefiting patients, providers, hospitals, and payers such as Medicare and private health insurance. Randomized, active-controlled clinical trials are required to compare the newer liposomal bupivacaine to continuous peripheral nerve blocks. The ultimate objective of the proposed research study is to determine if liposomal bupivacaine in a peripheral nerve block is at least non-inferior to a continuous peripheral nerve block following moderate-to-severely painful ankle surgery.

This is a single-center clinical trial. The investigators will randomize participants to either a liposomal bupivacaine combined with unencapsulated bupivacaine single-injection popliteal-sciatic and saphenous nerve block group, or single injections of unencapsulated bupivacaine followed by a continuous popliteal-sciatic bupivacaine infusion.

DETAILED DESCRIPTION:
For individuals of childbearing potential, a sample of urine will be collected before any study interventions to confirm a non-pregnant state (this is standard procedure for all surgical patients). Participants will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask and positioned prone. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area of insertion on the ipsilateral side as the surgery will be sterilely prepared, and a clear, sterile, fenestrated drape applied.

Treatment group allocation (randomization). Participants will be randomized and allocated to one of two possible treatments groups by the investigational pharmacist based on computer-generated lists in a 1:1 ratio stratified by treatment center and surgical procedure in blocks of 4. All study medication will be prepared and provided by the Investigational Drug Service and the syringes never shown to the participants or surgeons to retain masking (liposomal bupivacaine is white while unencapsulated bupivacaine is clear).

Treatment groups:

1. Experimental (includes liposomal bupivacaine)
2. Standard-of-Care (control)

Popliteal-sciatic nerve block. The sciatic nerve bifurcation will be identified by ultrasound in the short-axis view. The bifurcation will be defined as the most proximal point at which the tibial and common peroneal nerves have separated. Using ultrasound guidance, a standard Tuohy block needle will be advanced through a skin wheal of lidocaine until its tip is in the hypoechoic area immediately distal to the sciatic nerve bifurcation where the 2 branches of the sciatic nerve are adjacent but distinct deep to the paraneurium between the epineurium and paraneurium (the "subparaneural space/compartment"). Twenty milliliters of study fluid will be injected in divided doses with repeated negative aspiration. The study fluid will be comprised of:

Experimental Group: 10 mL of unencapsulated bupivacaine 0.375% and 10 mL of liposomal bupivacaine 1.33% (Exparel, Pacira BioSciences, Tampa, Florida) admixed within a 20 mL syringe.

Standard-of-Care Group: 20 mL of unencapsulated bupivacaine 0.375% with epinephrine (1:400,000) within a 20 mL syringe.

Perineural catheter insertion: The same needle will be redirected cephalad and inserted approximately 10 cm proximal superficial to the paraneurium ("supraparaneural" or "subepimyseal"). Normal saline will be injected to ensure there is no spread deep to the paraneurium and creating a pocket of fluid into which a perineural catheter will be advanced 3 cm past the needle tip. The needle will be removed and the catheter secured with surgical glue and an occlusive dressing. Using this protocol, the subsequent perineural infusion of study fluid will remain separated from the injectate deep to the paraneurium distal to the sciatic bifurcation to avoid a "washout" effect of the encapsulated and unencapsulated bupivacaine injected previously.

Adductor canal (saphenous) nerve block [standard-of-care]. Using ultrasound guidance, a standard Tuohy block needle will be used to anesthetize the saphenous nerve. Twenty milliliters of study fluid will be injected in divided doses with repeated negative aspiration. The study fluid will be comprised of:

Experimental Group [research specific]: 10 mL of unencapsulated bupivacaine 0.375% and 10 mL of liposomal bupivacaine 1.33% (Exparel, Pacira BioSciences, Tampa, Florida) admixed within a 20 mL syringe.

Standard-of-Care Group [standard-of-care]: 20 mL of unencapsulated bupivacaine 0.375% with epinephrine (1:400,000) within a 20 mL syringe.

A successful catheter insertion will be defined as sensory-block onset in all nerve distributions at the level of the ankle within the 30 minutes following the local anesthetic injection. In case of failure, the patient will be removed from further study.

Intraoperative protocol. Sedation or a general anesthetic will be permitted by the clinicians in the operating room who will be masked to treatment group assignment.

Postoperative protocol. As inpatients, our current standard analgesic protocol will be followed: acetaminophen 975-1000 mg po QID, oxycodone 5-10 mg po q4 h prn moderate pain (NRS 4-7), and morphine 1-2 mg IV prn severe pain (NRS>7). Prior to discharge, participants will all be provided with a prescription for oxycodone (5 mg tablets) by their surgeon, as dictated by our current standard of care. Prior to discharge from the recovery room a perineural infusion will be initiated (basal rate 5 mL/h; patient-controlled bolus of 4 mL; 30 minute lockout) with the reservoir (500 mL) and pump provided by the Investigational Drug Service and continued until postoperative day 3 or until the reservoir is exhausted. Contents of the reservoir will be determined by treatment group assignment:

Experimental Group [research specific]: normal saline.

Standard-of-Care Group [standard-of-care]: Unencapsulated bupivacaine.

On postoperative day 3 or when the reservoir is exhausted, participants themselves or their caretaker will remove the occlusive dressing and withdraw the catheter with gentle traction and rotation at home. The devices are single-use and disposable. Following study completion, the results will be mailed electronically or by the United States Postal Service to all enrolled participants in written form using non-technical (e.g., "layperson") language.

Outcome measurements. The investigators have selected outcome measures that have established reliability and validity, with minimal inter-rater discordance, and are recommended for pain clinical trials by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus statement.

Each time the end points are measured, participants will be instructed to respond for the previous 24 hours. The exception will be on Day 1 because at this time point, the interest is in participants' experiences subsequent to discharge from the recovery room. During this day only, participants will be instructed to respond for the period of time since they were discharged from the recovery room.

The investigators will record basic anthropomorphic characteristics (e.g., age, physiological sex, height, and weight), intervention characteristics (e.g., duration of application), surgical characteristics (e.g., surgical duration) and protocol deviations / adverse events. All data collection following the day of the intervention (Day 0) will be collected daily by telephone on postoperative days 1-7. Data will be collected by the investigators, Program Manager, and/or research coordinators specifically trained in these instruments' application, minimizing inter-rater discordance and standardizing responses. Observers masked to treatment group assignment will perform all postoperative assessments.

Primary outcome measure: The primary outcome measure will be a combination of daily "average" NRS and opioid consumption in oxycodone equivalents. In order to claim that Exparel is non-inferior to a perineural bupivacaine infusion for each postoperative day, both NRS and opioid consumption must be at least non-inferior for that day. The investigators will use a stepwise gatekeeping statistical procedure beginning on Day 1 and progressing daily through Day 7. Using this statistical method, no adjustment in alpha will be necessary to control Type 1 error through all 7 days.

Hypothesis 1: Following ankle surgery and single-injection unencapsulated bupivacaine popliteal-sciatic and saphenous nerve blocks, analgesia will be at least non-inferior in the 1st postoperative week with liposomal bupivacaine added to the initial nerve blocks compared with a 3-day popliteal-sciatic perineural unencapsulated bupivacaine infusion (daily average pain intensity as measured with the Numeric Rating Scale).

Current/present, worst, least, and average surgical limb pain will be assessed using a Numeric Rating Scale (NRS) as part of the Brief Pain Inventory (short form) on Days 1-3, and the "average" and "worst/maximum" NRS collected on postoperative days 4-7. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, zero equivalent to no pain and 10 equivalent to the worst imaginable pain. The NRS has been demonstrated to be a valid and reliable measure in multiple pain states and following analgesic interventions. In addition, NRS scores correlate well with other measures of pain intensity, and demonstrate high test-retest reliability in chronic nociceptive and neuropathic pain states. These NRS characteristics led to recent IMMPACT consensus recommendations for use of the 10-point NRS of pain intensity for pain trials.

Hypothesis 2: Following ankle surgery and single-injection unencapsulated bupivacaine popliteal-sciatic and saphenous nerve blocks, opioid consumption will be at least non-inferior in the 1st postoperative week with liposomal bupivacaine added to the initial nerve block compared with a 3-day perineural bupivacaine HCl infusion (as measured in daily cumulative oxycodone equivalents).

Opioid analgesic consumption in oxycodone equivalents will be recorded at all time points (Table 2), with a secondary outcome measure of high importance being the cumulative opioid dose in oral oxycodone equivalents for the first 7 postoperative days following recovery room discharge. The two treatment groups' daily opioid consumption will also be compared at all timepoints.

Additional Secondary Outcome Measures.

Brief Pain Inventory (Interference Subscale). It is well-recognized that, "pain is a complex, multidimensional, sensory, and emotional experience that is individually perceived and described in many different ways." This observation has led to consensus recommendations that "multiple core domains and related measures be considered in pain treatment trials," that "tap into a wider experience of pain over time and its impact on functioning and quality of life." Therefore, the proposed trial will include the Brief Pain Inventory, an instrument that includes-in addition to pain intensity scales-seven measures evaluating the pain's interference with physical and emotional functioning, such as sleep, relations with others, and enjoyment of life. It is this 7-question Interference Scale that will be applied on postoperative days 1-3. The Brief Pain Inventory has been used and validated in countless clinical pain-related studies. This instrument is associated with minimal participant burden and is easily interpreted by patients of all ages and education levels. It has high test-retest reliability and correlates well with much longer questionnaires, including the McGill measures and EuroQol.

In addition to the outcomes described above, The investigators will record awakenings due to pain at each data collection phone call with the two groups compared on the cumulative awakenings over the entire first postoperative week. The investigators will also record the day of discharge, side effects of the perineural infusion, and adverse events. The latter two are qualitative variables that cannot be ranked, and are thus exploratory in nature.

Sample Size Determination. The investigators will include 130 participants who received at least some of the perineural infusion within the analysis (10 additional for dropouts). This will be a non-inferiority study using 65 patients from one of Dr. Ilfeld's previously published clinical trials (PMID 26962712) to determine the sample size. These previous participants had single-injection sciatic-popliteal and adductor canal nerve blocks and a subsequent continuous popliteal-sciatic nerve block, as will the standard-of-care group of the proposed trial. On postoperative day 1 their mean (SD) pain intensity as measured with the numeric rating scale was 2.6 (2.1). While the exact magnitude of the minimal clinically important difference between two treatment groups remains unknown, the investigators propose a noninferiority margin = 1.0 as a conservative estimate.

The investigators simulated numeric rating scale for 10,000 trials by assuming normal distribution with mean 2.6 and standard deviation 2.1, then rounding to nearest integer in the range 0 to 10. Assuming no difference between groups, n=65 participants per group, the lower limit of 95% confidence interval associated with Wilcoxon Rank Sum test is greater than -1 (noninferiority margin) in 80% of the simulated trials. Similarly, opioid (oxycodone) consumption is expected to follow a truncated normal distribution with mean (SD) 10 mg (13 mg), and minimum value 0 mg. Simulated 10,000 trials under these assumptions, with only 25 participants per group, the lower limit of 95% confidence interval associated with Wilcoxon Rank Sum test is greater than -10 mg (noninferiority margin, again, a conservative value that will not be questioned by reviewers, editors, or readers) in 93% of the simulated trials. . Non-inferiority in both pain and opioid consumption will be required to claim overall non-inferiority for each postoperative day beginning the day after surgery and progressing through postoperative day 7; therefore, no adjustment in alpha is necessary to control Type 1 error. The investigators will include 130 participants who received at least some of the perineural infusion within the analysis (10 additional for dropouts). To allow for up to 10 dropouts, the investigators request a total of up to 140 participants.

General statistical approach. Baseline characteristics of the randomized groups will be summarized with means, standard deviations, and quartiles. Balance between groups will be assessed. Specifically, standardized differences will be calculated using Cohen's d whereby the difference in means or proportions is divided by the pooled standard deviation estimates. Any key variables (age, sex, height, weight, BMI, and surgical procedure) with an absolute standardized difference greater than 1.96×√(2/n) = 0.344, where n=65 is the target sample size per group, will be noted and included in a sensitivity analysis with a generalized linear model (e.g. ordinal regression for pain severity NRS or logistic regression for incidence rates) to obtain an estimate of the treatment effect adjusted for the imbalanced covariate(s). If key model assumptions are violated (i.e. homoscedasticity or Gaussian distribution for linear models), data transformations and/or alternative generalized linear models will be applied as appropriate. Missing data is expected to be negligible. In the event of unexpected missing data, multiple imputation by chained equations will be applied to obtain estimates of treatment effects under the assumption of missing at random. The imputation model will exhaustively consider all measured baseline covariates and longitudinal observations to maximize the likelihood that the missing at random assumption is met.

Analysis of the primary end point. All analyses will initially be for non-inferiority, followed by superiority testing if applicable. The primary analytic approach will be an unadjusted two-sample Mann-Whitney U test of the daily average NRS and opioid consumption in oxycodone equivalents for Days 1-7. If any key variables are imbalanced at baseline, a linear regression model, or appropriate generalized linear model, adjusting for those variables will be applied. In order to claim that liposomal bupivacaine is non-inferior to a perineural unencapsulated bupivacaine infusion for each postoperative day, both Hypotheses 1 and 2 must be at least non-inferior for that day. The investigators will use a stepwise gatekeeping statistical procedure beginning on Day 1 and progressing daily through Day 7. Using this statistical method, no adjustment in alpha will be necessary to control Type 1 error through all 7 days. The p-value and 95% confidence interval associated with the estimated group difference in average daily NRS will be provided. P<0.05 will be considered statistically significant.

Analysis of the secondary end points. All analyses will initially be for non-inferiority. Of note, testing for non-inferiority by comparing the limits of conventional two-sided 95% CIs to prespecified non-inferiority margins does not preclude the possibility of concluding inferiority or superiority if the same CI excludes zero. Continuous endpoints will be analyzed with the same approach as the primary endpoint. Binary endpoints will be analyzed with Fisher's Exact test for two proportions, or logistic regression in the event of imbalance on key baseline variables. Ordinal endpoints will be analyzed with the Armitage trend test, or cumulative link regression model, as warranted. Nominal 95% confidence intervals will be provided for secondary analyses.

Treatment effects will also be assessed at individual time points regardless of preceding results, and no adjustments will be made for testing multiplicity.

Secondary outcomes in descending order of importance (gatekeeping procedure) following the primary outcome (Days 1-7):

Gatekeeping order : Outcome Time Frame

1. Cumulative opioid use (oxycodone equivalents) Postop days 1-7
2. Median maximum NRS over entire study period Postop days 1-7
3. Cumulative awakenings due to pain Postop days 1-7
4. Daily Brief Pain Inventory interference subscale Postop days 1-3
5. Daily "worst" (maximal) NRS Postop days 1-7
6. Daily "least" (maximal) NRS Postop days 1-7
7. Side effects [qualitative only] Postop days 1-7
8. Adverse events [qualitative only] Postop days 1-7

Complications. The investigators will record all related complications. These complications cannot be "ranked", but rather the two groups will be compared descriptively on each of these possible adverse events.

No formal interim analyses are planned. Sub-group analyses based on BMI median split (2 sub-groups) and surgical procedure type will be conducted. Within each subgroup the approach described for the primary analysis will be repeated. For NRS for pain and opioid use on each postop day, the 95% confidence intervals associated with Wilcoxon Rank Sum test comparing treatment groups will be derived.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of at least 18 years of age
2. Undergoing a primary, unilateral, moderate-to-severely painful ankle surgery
3. Planned single-injection adductor canal nerve block and popliteal-sciatic catheter
4. Weight > 50 kg (to minimize the risk of local anesthetic toxicity)

Exclusion Criteria:

1. chronic opioid or tramadol use: daily oxycodone equivalents > 20 mg for > 4 weeks
2. neuro-muscular deficit of the surgical limb
3. moderate pain (NRS > 3) in an anatomic location other than the surgical site
4. surgery outside the sciatic and saphenous nerve distributions
5. history of opioid misuse
6. inability to communicate with the investigators
7. inability to contact the investigators during the treatment period, and vice versa (e.g., lack of telephone access)
8. incarceration
9. pregnancy
10. allergy to amide local anesthetics or other study medication
11. active lower extremity infection or other contraindications to a peripheral nerve catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-06-22 (Estimated); Study Completion 2027-06-22 (Estimated)

PRIMARY OUTCOMES:
First postoperative week daily average pain level | Postoperative days 1-7
  The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, zero equivalent to no pain and 10 equivalent to the worst imaginable pain. The primary outcome measure will be a combination of daily "average" NRS and opioid consumption in oxycodone equivalents. In order to claim that liposomal bupivacaine is non-inferior to a perineural bupivacaine infusion for each postoperative day, both NRS and opioid consumption must be at least non-inferior for that day. We will use a stepwise gatekeeping statistical procedure beginning on Day 1 and progressing daily through Day 7. Using this statistical method, no adjustment in alpha will be necessary to control Type 1 error through all 7 days.
First postoperative week cumulative opioid consumption | Postoperative days 1-7
  Cumulative opioid consumption from recovery room discharge through postoperative day 7 measured in oxycodone equivalents. The primary outcome measure will be a combination of daily "average" NRS and opioid consumption in oxycodone equivalents. In order to claim that liposomal bupivacaine is non-inferior to a perineural bupivacaine infusion for each postoperative day, both NRS and opioid consumption must be at least non-inferior for that day. We will use a stepwise gatekeeping statistical procedure beginning on Day 1 and progressing daily through Day 7. Using this statistical method, no adjustment in alpha will be necessary to control Type 1 error through all 7 days.

SECONDARY OUTCOMES:
Daily worst/maximum pain | Collected daily postoperative days 1-7
  Worst surgical limb pain will be assessed using a Numeric Rating Scale (NRS) as part of the Brief Pain Inventory (short form) on Days 1-3, and the "worst/maximum" NRS collected on postoperative days 4-7. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
Daily "average" pain | Collected daily postoperative days 1-7
  "Average" surgical limb pain will be assessed using a Numeric Rating Scale (NRS) as part of the Brief Pain Inventory (short form) on Days 1-3, and the "average" NRS collected on postoperative days 4-7. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
Daily lowest/minimal pain | Collected daily postoperative days 1-3
  The lowest daily surgical limb pain will be assessed using a Numeric Rating Scale (NRS) as part of the Brief Pain Inventory (short form) on Days 1-3. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
Daily "current" pain | Collected daily postoperative days 1-3
  The current daily surgical limb pain at the time of the data-collection phone call will be assessed using a Numeric Rating Scale (NRS) as part of the Brief Pain Inventory (short form) on Days 1-3. The NRS is a highly-sensitive measure of pain intensity with numbers ranging from 0 to 10, zero equivalent to no pain and 10 equivalent to the worst imaginable pain.
Daily opioid consumption | Collected daily postoperative days 1-7
  Cumulative opioid dose of the previous 24 hours measured in oral oxycodone equivalents.
Brief Pain Inventory, short form (Interference Subscale) | Collected daily postoperative days 1-3
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale;(2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale.
Awakenings due to pain | Collected daily postoperative days 1-7
  The number of times the patient awoke the previous night due to pain
Days hospitalized | Postoperative days 0-7
  Number of days from the intervention until the day of discharge measured in 1-day increments.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided